CLINICAL TRIAL: NCT05458843
Title: Renal Considerations in the Heat Stress and Hydration Recommendations (Aim 2)
Brief Title: Renal Considerations in the Heat Stress Recommendations (Aim2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Zachary J. Schlader, Associate Professor Kinesiology, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 15402
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Hot Weather; Adverse Effect; Kidney Dysfunction; Kidney Injury; Hyperthermia; Dehydration
MeSH Terms: conditions — Hyperthermia; Dehydration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid replacement (Experimental)
  Interventions: Procedure: Fluid replacement
- No fluid replacement (Sham Comparator)
  Interventions: Procedure: No fluid replacement

INTERVENTIONS:
Procedure: Fluid replacement — Participants will drink Gatorade Zero ad libitum, up to 1 cup every 15 minutes.
  Arms: Fluid replacement
Procedure: No fluid replacement — Participants will not be permitted to drink.
  Arms: No fluid replacement

SUMMARY:
An epidemic of chronic kidney disease is occurring in laborers who undertake physical work outdoors in hot conditions. The reason for this is largely unknown, but may be related to kidney dysfunction caused by increases in body temperature and dehydration that elicit oxidative stress and inflammation in the renal tubules. The purpose of this study is to determine whether hydration status modifies the development of renal oxidative stress and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-44 y old
* Body mass index ≤35.0 kg/m2
* Self-reported to be healthy

Exclusion Criteria:

* Not within defined age range
* Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2
* Body mass index >35.0 kg/m2
* Current or history of any renal disease, heart disease, stroke, immune or autoimmune disease, and/or gastrointestinal disease/surgery
* Hypertension during screening (systolic blood pressure >139 or diastolic blood pressure >89)
* Using medications that blunt the physiological response to exercise (e.g., beta blockers)
* Prescription medication with a known side effect of impaired temperature regulation or fluid balance (e.g., diuretics)
* Positive pregnancy test at any time during the study or breast feeding
* Current tobacco or electronic cigarette use or consistent use within the last 2 years
* Answered "Yes" to any question on Page 1 of the PAR-Q+.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Peak urinary thioredoxin | Through study completion, up to twelve weeks
  Marker of renal oxidative stress
Peak urinary MCP-1 | Through study completion, up to twelve weeks
  Marker of renal inflammation

SECONDARY OUTCOMES:
Peak urinary [IGFBP7 x TIMP-2] | Through study completion, up to twelve weeks
  Kidney injury marker
Renal artery blood velocity | Through study completion, up to twelve weeks
  Measure of kidney blood flow
Segmental artery blood velocity | Through study completion, up to twelve weeks
  Measure of kidney blood flow

OTHER OUTCOMES:
Core body temperature | Through study completion, up to twelve weeks
  Heat strain variable
Mean skin temperature | Through study completion, up to twelve weeks
  Heat strain variable
Oxygen uptake | Through study completion, up to twelve weeks
  Heat strain variable
Heart rate | Through study completion, up to twelve weeks
  Heat strain variable
Blood pressure | Through study completion, up to twelve weeks
  Heat strain variable
Percentage change in body weight | Through study completion, up to twelve weeks
  Hydration status variable
Blood and plasma volume | Through study completion, up to twelve weeks
  Hydration status variable
Plasma osmolality | Through study completion, up to twelve weeks
  Hydration status variable
Urine osmolality | Through study completion, up to twelve weeks
  Hydration status variable
Urine specific gravity | Through study completion, up to twelve weeks
  Hydration status variable
Creatinine clearance | Through study completion, up to twelve weeks
  kidney function variable

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health, Bloomington, Indiana, United States